CLINICAL TRIAL: NCT05230940
Title: Multicenter,Randomized,Observational Blind Phase IIB Clinical Trial to Evaluate the Effectiveness,Immunogenicity and Safety of Two Doses of CoronaVac (Sinovac) Vaccine Against Two Doses of Inactivated COVID-19 Vaccine (TURKOVAC) in Healthy Adolescent (12-18 Years) Subjects
Brief Title: Efficacy, Immunogenicity, and Safety of TURKOVAC Vaccine Versus the CoronaVac Vaccine Against COVID-19 in Healthy Adolescent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TSB-VAC-COV-TUR-EF2B.06
Record Dates: First submitted 2022-02-05; First posted 2022-02-09 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Sars-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Vaccine; Efficacy; Immunogenicity; Safety; Adolescent
MeSH Terms: conditions — COVID-19 | interventions — TURKOVAC; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Multi-Centered, Randomized, National, Observer-blinded, Active-controlled, Phase IIB
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the study nurse is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TURKOVAC (Experimental): The dose of the TURKOVAC vaccine will be 3 μg/0.5 mL. It will be administered by injection to the left deltoid muscle of the upper arm, two doses are given 28 days apart.
  Interventions: Biological: TURKOVAC
- CoronaVac (Active Comparator): The dose of the CoronaVac vaccine will be 3 μg/0.5 mL. It will be administered by injection to the left deltoid muscle of the upper arm, two doses are given 28 days apart.
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: TURKOVAC — Inactive COVID-19 Vaccine - TURKOVAC
  Arms: TURKOVAC
Biological: CoronaVac — It has 600 subunit of SARS-CoV-2 virus antigen
  Arms: CoronaVac

SUMMARY:
This study is a multi-center, randomized, national, observer-blinded, active-controlled phase IIB clinical trial to determine the efficacy, immunogenicity, and safety of two-doses of inactive COVID-19 vaccine (TURKOVAC) vaccine versus the two-doses CoronaVac (Sinovac) vaccine in healthy adolescents aged 12-18 years.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the clinical efficacy of two-doses of TURKOVAC and two-doses of CoronaVac vaccines against symptomatic COVID-19 disease confirmed by real time-polymerase chain reaction (RT-PCR) in adolescents (12-18 years of age).

After the second dose of vaccine administration, the immunological responses of TURKOVAC and CoronaVac vaccines will be demonstrated by neutralizing antibodies and anti-spiked antibodies.

A total of 644 subjects will be enrolled. Subjects will be assigned according to randomization (1:1) for 2 different arms. The assigned vaccine will be administered to subjects in two doses on days 0 and 28.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be enrolled in this study:

1. Subjects who can voluntarily consent to participate in the study with their parents or legal representatives,
2. Subjects agreed to comply with all study visits and procedures (consented to give blood sample and nasopharyngeal swab, and receiving automated telephone calls from the study site),
3. No history of SARS-CoV-2 (within the last 12 months),
4. Consent of sexually active females to use effective contraception during the study,
5. Adolescent males or females who were at least 12 years old and not older than 18 years of age on the date of the informed consent signature,
6. In the opinion of the investigator, subjects who can comply with the study protocol during the study,
7. According to the vaccination program of the Ministry of Health, meeting the criteria for vaccination however, who voluntarily choose not to be vaccinated when rights are granted and subjects who agreed to receive one of the vaccines to be used in this study,
8. Not participating in another clinical trial.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Is acutely ill or febrile within 48 hours before or use of antipyretic or analgesic medication within 24 hours before planned administration of study vaccine. (Fever is defined as a body temperature is 38.0 °C. Subjects with mild illness and fever may be enrolled in the study at the discretion of the investigator),
2. Those who have used more than a single dose of Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) in the last 24 hours for a reason other than fever,
3. Subjects who are pregnancy or breastfeeding plan within (at least) 1 year following the second dose of vaccine,
4. Those with a history of SARS-CoV-2 (within the last 12 months),
5. Individuals with a current positive (PCR-based viral RNA detection) or past positive (serological testing or PCR-based viral RNA detection) diagnostic test result for SARS-CoV-2 infection,
6. Prior administration of an investigational or approved coronavirus (SARS-CoV, SARS-CoV-2, MERS-CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19,
7. Subjects with a history of cardiac diseases (cardiovascular disease, serious arrythmia, coronary artery disease, heart failure, cardiomyopathies, pulmonary hypertension etc.),
8. Subjects with uncontrolled hypertension,
9. Subjects with a first-degree relative with a history of coronary artery disease at an early age (presence of coronary artery disease before 55 years of age in males and 65 years of age in females),
10. Subjects with morbid obesity (Body Mass Index (BMI) ≥ 40),
11. Subjects with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and autoimmune bullous diseases,
12. Subjects with history of severe allergic reaction (i.e., anaphylaxis, generalized urticaria, angioedema, or other significant reaction) to any licensed or investigational vaccine or to any of the constituents of CoronaVac or TURKOVAC,
13. Subjects who have bleeding disorder considered a contraindication to intramuscular injection or phlebotomy,
14. Subjects who have immunosuppressive or immunodeficiency state (including HIV), asplenia, recurrent severe infections,
15. Subjects who received or planned to receive a licensed, live replicating vaccine (any vaccine other than the COVID-19 vaccine) within 28 days before or after the first study vaccination or a licensed inactivated or nonreplicating vaccine (any vaccine other than the COVID-19 vaccine) within 14 days before or after first study vaccination,
16. Subjects who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, within 6 months prior to screening, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study vaccine administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted,
17. To be using an immunostimulant, immune-modifying supplementary drug or herbal product or to have used it in the last month,
18. Subjects who have received systemic immunoglobulin or blood products in the past 12 months, or who plan to receive such products during the study,
19. Investigator, site coordinators, employees of TUSEB or the Clinical Research Organization (CRO) directly involved in the conduct of the study, or site staff members otherwise supervised by the Investigator or immediate family members of any of the previously mentioned individuals.
20. Subjects who have previously received any COVID-19 vaccines.

Exclusion criteria for the second dose of vaccine:

1. Before the second vaccination, in the case of an unresolved acute illness or in the acute phase of a chronic illness, the investigator should exclude COVID-19 and assess if the acute disease can recover in a short term.
2. If there is an adverse event after the first dose or newly occurred non-compliance with the inclusion/exclusion criteria which will be assessed by the investigator whether the study subjects can continue or not.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
COVID-19 Positivity Rate | 14 days after the second dose of vaccination
  The rate of positivity in a polymerase chain reaction (PCR) sample taken within 24 or 48 hours in subjects (symptomatic subject) with fever and other COVID-19 symptoms 14 days after the second vaccination dose.

SECONDARY OUTCOMES:
Protection Rates of TURKOVAC and CoronaVac Vaccines Against Symptomatic COVID-19 | 14 days after first dose of vaccination
  Protection rates of TURKOVAC and CoronaVac vaccines against symptomatic COVID-19 confirmed by real time-polymerase chain reaction (RT-PCR), 14 days after first dose of vaccination.
Protection rates of TURKOVAC and CoronaVac Vaccines Against Symptomatic COVID-19 | 14 days after second dose of vaccination
  Protection rates of TURKOVAC and CoronaVac vaccines against symptomatic COVID-19 confirmed by real time-polymerase chain reaction (RT-PCR), 14 days after second dose of vaccination.
The Protection Rates of TURKOVAC and CoronaVac Vaccines in Preventing Hospitalization and Death Against Severe COVID-19 | 14 days after second dose of vaccination
  The protection rates of two-doses of TURKOVAC and CoronaVac vaccines in preventing hospitalization and death against severe COVID-19 disease confirmed by real time-polymerase chain reaction (RT-PCR), 14 days after the second dose of vaccination.
The Incidence of Adverse Events (AEs) | Up to 30 minutes each dose of vaccination
  The incidence of adverse events (AEs) within after up to 30 minutes each dose of vaccination.
The Incidence of Undesirable Adverse Event | First day of vaccination to the following year after the last dose of vaccination
  The incidence of an undesirable adverse event from the first day of vaccination to the following year after the last dose of vaccination.
The Incidence of Undesirable Adverse Event | 7 days after each vaccination dose
  The incidence of undesirable adverse events within 7 days after each vaccination dose.
The Incidence of Serious Undesirable Adverse Events | 1 year after first and second dose vaccination
  The incidence of serious undesirable adverse events up to one year after first and second dose vaccination.
The Seropositivity Rate of SARS-CoV2 Specific Binding Antibody | 42, 56, 70, 126, 168, and 224 days after the first dose of vaccination
  The seropositivity rate of SARS-CoV2 specific binding antibody at 42, 56, 70, 126, 168, and 224 days after the first dose of TURKOVAC and CoronaVac vaccination.
  * The change in the geometric mean concentration (GMC) SARS-CoV2 anti-spike protein immunoglobulin G in the 42nd and 56th day compared to the baseline is 2 times.
Evaluation of SARS-CoV2 Neutralizing Antibodies | 42, 56, 70, 126, 168, and 224 days after the first dose of vaccination
  To evaluate SARS-CoV2 neutralizing antibodies by neutralization test at 42, 56, 70, 126, 168, and 224 days after the first dose of TURKOVAC and CoronaVac vaccination.
  * The change in the geometric mean concentration (GMC) and geometric mean titer (GMT) SARS-CoV2 neutralizing antibodies in the 42nd and 56th day compared to the baseline is 2 times.
T-Cell Evaluation | 70, 126, and 224 days after the first dose of vaccination
  To evaluate the SARS-CoV2 protein-peptide pool-specific T cells (T cell activation) on the first dose day and at 70, 126, and 224 days after the first dose. Geometric mean percentage (minimum 25 percent, maximum 75 percent) of SARS-CoV2 protein-peptide pool-specific T-cell determined by flow cytometry.
  * The success criterion for T cell activation is defined as the appearance of an anamnestic response.
The Incidence of Local and Systemic Signs and Symptoms | Through study completion, an average of 1 year
  The incidence of local and systemic signs and symptoms in TURKOVAC and CoronaVac vaccines will be evaluated with the chi-square test when the chi-square condition is provided, and the Fisher Exact Test when the chi-square condition is not provided.

CONTACTS AND LOCATIONS:
Overall Officials: Aslınur Özkaya Parlakay, Prof., Principal Investigator — Faculty Member
Locations (14):
- Turkey (Türkiye) (14):
  - Health Sciences University Adana City Training and Research Hospital, Pediatric Health and Diseases, Adana
  - Çukurova University Faculty of Medicine Department of Pediatric Infectious Diseases, Adana
  - T.R. Ministry of Health Ankara City Hospital, Pediatric Infectious Diseases Clinic, Ankara
  - Ankara University Faculty of Medicine Department of Pediatric Infectious Diseases, Ankara
  - Hacettepe University Faculty of Medicine Department of Child Health and Diseases Department of Pediatric Infectious Diseases, Ankara
  - Eskişehir Osmangazi University Faculty of Medicine, Department of Child Health and Diseases, Eskişehir
  - İstanbul University İstanbul Faculty of Medicine, Department of Pediatric Infectious Diseases, Istanbul
  - Marmara University Istanbul Pendik Training and Research Hospital, Pediatric Infectious Diseases Clinic, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşçıoğlu City Hospital, Pediatric Infectious Diseases Clinic, Istanbul
  - University of Health Sciences İstanbul Şisli Hamidiye Etfal Training and Research Hospital, Pediatric Infectious Diseases Clinic, Istanbul
  - Ege University Faculty of Medicine, Department of Child Health and Diseases, Izmir
  - T.R. Ministry of Health İzmir Provincial Health Directorate İzmir Health Sciences University Tepecik Training and Research Hospital, Clinic of Child Health and Diseases, Izmir
  - University of Health Sciences İzmir Dr. Behçet Uz Child Disease and Pediatric Surgery Training and Research Hospital, Izmir
  - Erciyes University Faculty of Medicine Department of Pediatric Infectious Diseases, Kayseri